CLINICAL TRIAL: NCT03715374
Title: Treatment of Periodontal Intrabony Defects With Platelet-Rich Fibrin and Anorganic Bovine Bone vs Collagen Membrane and Anorganic Bovine Bone. A Non-Inferiority Trial
Brief Title: Platelet-Rich Fibrin and Anorganic Bovine Bone vs Collagen Membrane and Anorganic Bovine Bone in Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, professor and chairman, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19102018
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Periodontal Attachment Loss; Periodontal Bone Loss; Periodontal Diseases
Keywords: Platelet rich fibrin; bone graft; non inferiority trial
MeSH Terms: conditions — Periodontal Attachment Loss; Alveolar Bone Loss; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF+ABB treated patients (Experimental): Periodontal surgery with Platelet Rich Fibrin is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Anorganic bovine bone material will be applied to the entire root surfaces ; then, A prf membrane is positioned above the filling material. Finally the flap will be positionated and sutures completed by interrupted sutures.
  Interventions: Procedure: Periodontal Surgery with PRF+ABB
- Collagen Membrane + ABB treated patients (Active Comparator): Periodontal surgery with collagen membrane is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Anorganic bovine bone material will be applied to the entire root surfaces ; then, A collagen membrane is positioned above the filling material. Finally the flap will be positionated and sutures completed by interrupted sutures.
  Interventions: Procedure: Periodontal Surgery with Collagen Membrane +ABB

INTERVENTIONS:
Procedure: Periodontal Surgery with PRF+ABB — Patients will be treated by periodontal surgical flaps with the addition of PRF+ Anorganic Bovine Bone filling material
  Arms: PRF+ABB treated patients
Procedure: Periodontal Surgery with Collagen Membrane +ABB — Patients will be treated by periodontal surgical flaps with the addition of Collagen Membrane + Anorganic Bovine Bone filling material
  Arms: Collagen Membrane + ABB treated patients

SUMMARY:
The primary outcome of periodontal reconstructive therapy is to regenerate all tissues of the periodontium including a functional periodontal ligament, alveolar bone and cementum. A number of treatment modalities including the use of bone grafts, guided tissue regeneration (GTR), and the addition of biological agents have been used with large heterogeneity in the clinical and histological outcomes. The rationale of using a filling material when treating unfavorable and large intrabony defects (IBDs) with membranes or biological agents consists of sustaining the overlying soft tissues in the presence of a non-contained defect's architecture, at the same time enhancing the stability of coagulum; and facilitating the proliferation of mesenchymal progenitor cells. Among bone grafts available, anorganic bone bone (ABB) have been widely used in periodontics for the treatment of IBDs In recent years, the increasing understanding of the role of growth factors (GFs) in the wound healing process suggested the use of these biological agents in the regenerative treatment of periodontal bony defects. Noninferiority trials are designed to demonstrate that the effect of a new treatment is adequately similar to an active control by more than a specified margin The aim of this study is to verify if the combined use of PRF (Platelet Rich Fibrin) and ABB in the management of IBDs may be a treatment modality that is clinically "not inferior" compared to the membrane + ABB one, since the combined periodontal regenerative technique has been already tested in literature as a "gold standard" periodontal regenerative technique.

DETAILED DESCRIPTION:
Experimental Design This is a prospective, randomized and controlled clinical trial designed to evaluate the clinical and radiographic outcomes 12 months after two treatment modalities of IBDs: test sites ( TS) will be treated by a combination of PRF and ABB; control sites (CS) will receive the combined treatment of collagen membrane + ABB. The patients enrolled will exhibit unfavorable IBDs and all experimental sites will be accessed with a simplified papilla preservation flap (SPPF) procedure. The filling material (ABB) will be common to both treatments: therefore, the investigation focused on the addictive effect of PRF used instead of COLLAGEN MEMBRANE. Collagen membrane is chosen as the active control (AC) as it is currently considered as the "gold standard" among the biological agents for the treatment of IBDs.

A non-inferiority trial (NIT) is designed to verify whether to use PRF instead of collagen membrane in association with ABB can lead to not inferior therapeutic results, reducing the treatment's cost and allowing the clinicians to use autogenous materials only.

Study Population 62 patients (33 males and 29 females) aged 42 to 64 years (mean: 53±12) seeking treatment at the Unit of Periodontology of the "G. D'Annunzio" University of Chieti- Pescara, Italy, and affected by moderate-to-severe chronic periodontitis, will be selected for the study. The inclusion criteria are: 1) no systemic diseases; 2) no medications affecting periodontal status during the previous 6 months; 3) not pregnant or lactating; 4) non-smoker; and 5) the following dental and periodontal factors: a full-mouth plaque score (FMPS)25 and a full-mouth bleeding score (FMBS)26 < 20% at the time of surgery, no periodontal therapy in the 2 previous years, no inadequate endodontic treatment at the experimental sites, no dental mobility, ≥ 20 teeth, exhibit vertical bone loss detected by radiographic examination ( ACL (alveolar crest level) - (BD bottom of the defect) distance = BDD (Bone defect depth ) ≥ 4 mm and a probing pocket depth (PPD) ≥ 5mm when evaluated 12 weeks after non- surgical therapy [ scaling and root planing ( SRP)]. Only predominantly 1-, combined 1- and 2-, 2-walls defects or teeth with a defect angle ≥ 36° were considered in this study (unfavorable IBDs). To be included in this category, the IBDs should not have a 3-wall component >20% of the total defect depth. The architecture of the defect had to be confirmed by observation during the surgical intervention. Each patient will participate in the study with a single experimental site. In the case that a patient will have more than one IBD with clinical features that could be eligible for study, the most severe defect will be chosen. The participants volunteered for the study after they will receive verbal and written information and signed a consent form approved by the Ethical Committee of the G. D'Annunzio University of Chieti - medical faculty. The study protocol is in accordance with the Declaration of Helsinki of 1975, revised in Tokyo in 2004. The study was performed from February 2013 to December 2016. Four months before the surgical treatment, all 44 patients will undergo SRP by ultrasonic instruments II and hand curettes¶ and motivational instructions on oral home care.

ELIGIBILITY:
Inclusion Criteria:

* a full-mouth plaque score (FMPS) 25 and a full-mouth bleeding score (FMBS) 26 < 20% at the time of surgery
* to have at least 20 teeth,;
* at least 1 tooth exhibiting vertical bone loss detected by radiographic examination (alveolar crest level [ ACL]
* bottom of the defect [ BD] distance = Bone defect depth [ BDD]) ≥ 4 mm and a probing pocket depth (PPD) ≥ 5mm when evaluated 12 weeks after phase I non- surgical therapy [ scaling and root planing ( SRP)].

Exclusion Criteria:

* no systemic diseases
* no medications affecting periodontal status during the previous 6 months
* not pregnant or lactating;
* non-smoker
* no periodontal therapy in the 2 previous years,
* no inadequate endodontic treatment, no dental mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Periodontal attachment gain | 1 year
  Reduction of the distance between the cementum-enamel junction and the depth of the probable site

SECONDARY OUTCOMES:
Bone gain | 1 year
  Gain of bone into the periodontal defects

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided